CLINICAL TRIAL: NCT06133335
Title: Prevalence of Periodontal Disease in Adult Patients Suffering From Cystic Fibrosis in the University Hospital of Reims: a Pilot Study
Brief Title: Cystic Fibrosis and Periodontal Diseases
Acronym: MucoParo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO23074
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis; Periodontitis; Gingivitis
Keywords: Cystic fibrosis; Periodontitis; gingivitis
MeSH Terms: conditions — Cystic Fibrosis; Periodontitis; Gingivitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cystic fibrosis subjects (Other): Adult patients with cystic fibrosis consulting the Resource and Competence Center for Cystic Fibrosis at the C.H.U. from Reims
  Interventions: Other: Periodontal examination

INTERVENTIONS:
Other: Periodontal examination — Periodontal examination is performed using PCP UNC15 periodontal probe (common diagnostic method not added by research).
  Gingival smear from various points in the oral cavity. This intervention consists in a smear of gingival area with an absorbent paper point into the space between the gum and the tooth (Jourdain et al. 2018). The objective of this technique is to remove the various elements of the periodontal pocket and in particular the desquamated cells.

SUMMARY:
The number of CF adults is increasing year after year (61.7% in 2021) confirming that patients are living longer. These data do not leave aside the desire to see CF patients "age well" considering of all the comorbidities linked to aging.

Among these comorbidities, the oral repercussions of cystic fibrosis and its treatments remain to this day little investigated. We know, however, that oral health, and periodontal health, is closely linked to general health. Indeed, the oral cavity presents one of the richest microbiota in the body, made up of bacteria, viruses, yeasts and archae organized into a biofilm at the interface of periodontal tissues. Periodontal diseases are partly linked to an imbalance in and loss of diversity within the commensal periodontal flora, aggravated by risk factors such as diabetes, which affects many CF adults. Early detection and treatment of periodontal diseases are therefore of primary interest in patients at increased risk of respiratory infections such as CF patients. This transversal research project aims to study the oral repercussions, notably periodontal disease prevalence in cystic fibrosis (CF) adult patients.

Thus, this program will allow, on the one hand, the acquisition of clinical and biological data on periodontal and/or dental pathologies from which adult CF patients may suffer. These data will be accessible through an oral and periodontal clinical examination that will allow the identification of diagnostic clues. The quality of life related to oral health will also be investigated using a self-administered questionnaire. Clinical and biological data commonly recorded in the context of the medical follow-up of CF patients (ventilatory capacity, glycemic status, cytobacteriological examination of sputum, etc.) will also be taken into account in order to study any correlations with periodontal status.

On the other hand, on a more fundamental level, this work aims to investigate the impact of CFTR protein dysfunction on the local immunity of the oral cavity and more particularly on the expression of antimicrobial peptides at the level of the periodontium.

Thus this project is articulated around a strong axis which is "aging well" for adult CF patients thanks to the improvement of knowledge and ultimately the prevention of comorbidities linked to aging in CF adult patients and particularly those related to oral health.

DETAILED DESCRIPTION:
The main objective of this study is to determine the prevalence of periodontal disease in adult CF subjects followed at CRCM of the CHU of Reims. Periodontal diseases (periodontitis and gingivitis) will be diagnosed according to the international classification of periodontal diseases (Chicago 2017). Periodontal examination will be performed with periodontal probe PCP UNC15. The diagnosis of periodontal disease is defined from the decision algorithm including measurement of interdental attachment loss (CAL), measurement of gingival recession (REC) and depth of vestibular or lingual pocket (PPD) (Tonetti and Sanz 2019).The clinical indices noted will therefore include: pocket depth on probing, gingival recession (Ramfjord 1959), periodontal attachment loss (CAL=PPD+REC) and bleeding index (BOP) (Ainamo and Bay 1975).

The secondary objectives are:

1. To Investigate an association between the presence of periodontal disease and:

   * the CFTR expression genotype (type of mutation)
   * the ventilatory capacity (FEV1)
   * the treatments administered and their mode of administration
   * the value of glycated hemoglobin (Hba1c%)
2. To assess the prevalence of carious lesions in adult cystic fibrosis patients
3. To assess the impact of cystic fibrosis and its treatments on oral health-related quality of life.
4. To look for an association between periodontal clinical indices and the level of expression of genes encoding antimicrobial peptides

ELIGIBILITY:
inclusion criteria :

* Adult patients affected by cystic fibrosis consulting the Resource and Competence Center for Cystic Fibrosis of the C.H.U. from Reims
* Patient who signed the consent
* Patient affiliated to the French social security system

exclusion criteria :

* A medical history that could compromise the protocol (psychiatric, medical disorders)
* Cancer
* Pregnancy
* Patients protected by law, minors, adults under guardianship and curatorship, people hospitalized without their consent and not protected by law, or people deprived of their liberty

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periodontal disease | Day 0
  Periodontal Disease will be diagnosed according to the new classification of periodontal diseases (Chicago, 2017) and defined by the decision-making algorithms (Tonetti and Sanz, 2019). Diagnosis will be based on Buccal or lingual Clinical attachment level (CAL), Recession (REC) and Periodontal Pocket Depths (PPD) measurement.

SECONDARY OUTCOMES:
Oral Health Quality of Life | Day 0
  GOHAI validated in French for general population -Tubert-Jeanin et al., 2003)
Prevalence of carious lesions | Day 0
  Evaluated by ICDAS (International Caries Detection and Assessment Score) (Ismaïl et al., 2007)
Level of expression of antimicrobial peptides genes | Day 0
  Evaluated by ΔΔCt compared to a classically used reference gene

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France